CLINICAL TRIAL: NCT07113808
Title: Clinical Medical Quality Control Management of Pediatric Intravenous Contrast-Enhanced Ultrasound(CEUS) in China: A Multi-Center Study
Brief Title: Pediatric Intravenous Contrast-Enhanced Ultrasound(CEUS) in China
Acronym: CEUS
Status: Recruiting | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Shenzhen Children's Hospital (Other Government); Children's Hospital of Chongqing Medical University (Other); Tianjin Children's Hospital (Other); Kunming Children's Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); West China Hospital (Other); Yuying Children's Hospital of Wenzhou Medical University (Other); Xian Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Jingjing Ye, Director of the Ultrasound Department, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: JiYe
Record Dates: First submitted 2025-07-17; First posted 2025-08-11 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Neoplasm; Abdominal Injury; Ascites
MeSH Terms: conditions — Abdominal Neoplasms; Abdominal Injuries; Ascites | interventions — contrast agent BR1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: contrast-enhanced ultrasound examination — to evaluate the the application of contrast-enhanced ultrasound examination in children with intra-abdominal diseases that require clear diagnoses aged from 29 days to 18 years old
Drug: SonoVue® — perform contrast enhanced ultrasound (CEUS) using Sonovue as the contrast agent

SUMMARY:
The goal of this clinical trial is to evaluate the application of intravenous contrast-enhanced ultrasound examination in children with intra-abdominal diseases that require clear diagnoses. The main questions it aims to answer are:

* Is intravenous contrast-enhanced ultrasound helpful for the diagnosis of intra-abdominal diseases in children?
* What medical problems do participants have when participating in intravenous contrast-enhanced ultrasound examination?
* How can ultrasound doctors conduct intravenous contrast-enhanced ultrasound examinations in a standardized manner? Researchers will performing intravenous contrast-enhanced ultrasound examinations on participants and collecting research subjects to establish a multicenter clinical data database.

Participants will:

* Perform abdominal ultrasound examination to assess the condition.
* At least conduct one intravenous contrast-enhanced ultrasound examination. Based on the result of the contrast examination, decide whether to conduct another examination.
* Keep a diary of their symptoms and therapeutic process in 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 29 days to 18 years old;
2. The clinical diagnosis was abdominal space-occupying lesions, blunt abdominal trauma, ascites of unknown cause, and children with suspected abdominal disease but other examinations could not identify the cause.

Exclusion Criteria:

1. Allergic to sulfur hexafluoride or other components;
2. Heart disease with right-to-left shunt/severe pulmonary hypertension /uncontrolled systemic hypertension/respiratory failure/heart failure/severe arrhythmia;
3. Electrocardiogram, echocardiography or clinical manifestations of myocardial ischemia;
4. Patients with severe blood system diseases or infectious diseases;
5. Hypercoagulable state and recent history of thrombosis;
6. Severe hepatic and renal insufficiency;
7. Patients with respiratory tract infection or congenital respiratory malformation.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients in Children's Hospital Affiliated to Zhejiang University School of Medicine, Second Affiliated Hospital of Zhejiang University School of Medicine, Shenzhen Children's Hospital, West China Hospital of Sichuan University, Children's Hospital of Chongqing Medical University, Tianjin Children's Hospital, Xi 'an Children's Hospital, Yuying Children's Hospital Affiliated to Wenzhou Medical University, Kunming Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity | Thirty days after the last venous ultrasound contrast examination
  to calculate the sensitivity of venous contrast-enhanced ultrasound examination in children
specificity | Thirty days after the last venous ultrasound contrast examination
  to calculate the specificity of venous contrast-enhanced ultrasound examination in children
Positive predictive value | Thirty days after the last venous ultrasound contrast examination
  to calculate the positive predictive value of venous contrast-enhanced ultrasound examination in children
Negative predictive value | Thirty days after the last venous ultrasound contrast examination
  to calculate the negative predictive value of venous contrast-enhanced ultrasound examination in children

OTHER OUTCOMES:
adverse event rate | Thirty days after the last venous ultrasound contrast examination
  to calculate the adverse event rate of venous contrast-enhanced ultrasound examination in children

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes